CLINICAL TRIAL: NCT04573023
Title: A Phase III Study of JR-141 in Patients With Mucopolysaccharidosis II (STARLIGHT)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JR-141-GS31
Record Dates: First submitted 2020-09-17; First posted 2020-10-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II | interventions — idursulfase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- JR-141 2.0 mg/kg/week (Experimental)
  Interventions: Drug: JR-141
- administered as the standard of care: idursulfase (ELAPRASE®) (Other): standard of care-controlled study
  Interventions: Drug: Idursulfase
- Rescue arm (Other)
  Interventions: Drug: JR-141 or Idursulfase

INTERVENTIONS:
Drug: JR-141 — IV infusion, 2.0 mg/kg/week
  Arms: JR-141 2.0 mg/kg/week
Drug: Idursulfase — IV infusion
  Arms: administered as the standard of care: idursulfase (ELAPRASE®)
Drug: JR-141 or Idursulfase — The subjects who have achieved the pre-specified criteria* are able to change the drug.
  *If a subject in Idursulfase group shows decline in their neurocognitive outcome, idursulfase can be switched to JR-141.
  If a subject in JR-141 group shows decline in their peripheral outcome, JR-141 will be switched to idursulfase.
  Arms: Rescue arm

SUMMARY:
A Global Phase III multicenter, randomized, assessor-blinded, active-controlled designed to evaluate safety and efficacy of study drug for the treatment of the MPS II.

ELIGIBILITY:
Inclusion Criteria:

* A patient who voluntarily signs an Institutional Review Board or Independent Ethics Committee-approved written informed consent form. If the patient is aged under 18 years (aged under 16 years in the UK) at the time of enrollment or willingness to participate in the study cannot be confirmed due to MPS II-related intellectual disability, the patient's legally acceptable representative (e.g., his/her parents or guardians) may sign the informed consent on behalf of the patient. Written informed assent should be obtained from the patient, wherever possible.
* Patients with confirmed diagnosis of MPS II
* Naïve patients or patients who are receiving stable enzyme replacement therapy with idursulfase for more than 12 weeks before starting administration of JR-141 or idursulfase for this study.
* Patients or patients whose partners are of child-bearing potential agree to use a medically accepted, highly effective method of contraception being use of condoms from the time of informed consent.

<Cohort A>

* Patients aged 36-42 months old at the time of ICF signing: patients must have a standard score measured by the BSID-III of 85 or less at screening.
* Patients aged 43-71 months old at the time of ICF signing: patients must EITHER have (1) A DQ measured by BSID-III of 20 to 85 at screening OR (2) A composite standard score on NVI measured by KABC-II of 85 or less at screening (only who can perform KABC-II)
* Patients aged 30-35 months old at the time of randomization and who are judged as having the severe phenotype by the Expert Board.

<Cohort B>

* Patients 6 years of age or older at the time of ICF signing and whose IQ are 70 and higher.
* Enrollment of subjects in Cohort B is contingent on the availability in that country of a validated country-specific version of the test (either WISC-V, WAIS-IV, or T.O.V.A.).
* Attenuated patients with 1 SD deficiency in the omission errors or variability domains of the T.O.V.A..
* Patients or patients whose female partners are of child-bearing potential i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile, agree to use a medically accepted, highly effective method of contraception, from the time of informed consent. The method of contraception must be used during the study until 90 days for male subjects, and 30 days for female subjects after the final study intervention administration.
* For subjects with hearing impairment requiring hearing aid(s), every effort has been made to encourage compliance with the use of functioning hearing aid(s) before baseline neurocognitive assessments, and parent/legally acceptable representative or subject agrees to encourage wearing them during the study and on neurocognitive testing days.

Exclusion Criteria:

* A patient with a history of HSCT with successful engraftment.
* A patient who has received gene therapy treatment at any point.
* A patient who is judged by the principal investigator or sub-investigator as being unable to undergo lumbar puncture, including those who have difficulties in taking position for lumbar puncture due to joint contracture or those who are likely to experience breathing difficulties during the lumbar puncture process.
* A patient who is enrolled in another clinical study that involves clinical investigations or use of any investigational product (drug or device) within 4 months before obtaining informed consent.
* Unable to comply with the protocol as determined by the principal investigator or subinvestigator.
* Judged by the principal investigator or subinvestigator to be ineligible to participate in the study due to a history of serious drug allergy or sensitivity including anesthesia or hypersensitivity to any component of JR-141.
* A patient who has a known or suspected local or general infection or is at risk of abnormal bleeding due to medical conditions or therapies.
* A patient who has documented mutation of other genes, including loci adjacent to the IDS gene that are known to be associated with developmental delay, seizures, or other significant CNS disorders.
* A patient who has documented loss of activity of sulfatases other than IDS.
* A patient who has had a ventriculoperitoneal shunt placed or any other brain surgery, or has a clinically significant ventriculoperitoneal shunt malfunction within 30 days of screening.
* A patient who is full time employee of the sponsor or research site personnel directly affiliated with this study or their immediate family members.
* A patient who otherwise is judged by the principle investigator or sub-investigator to be ineligible to participate in the study.
* The subject has a positive pregnancy test or is breastfeeding at screening or randomization.

[Only in France]

* Persons deprived of their liberty by a judicial or administrative decision, according to article L.1121-6 the Public Health Code (Code de la santé publique), adults who are the subject of a measure of legal protection or unable to express their consent according to article L. 1121-8 of the Code de la santé publique)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in levels of cerebrospinal fluid heparan sulfate from baseline (Cohort A) | Baseline to Week 53
Change in the raw scores of cognitive testing measured from baseline (BSID-III) (Cohort A) | Baseline to Week 105

SECONDARY OUTCOMES:
For regions other than US: Change in the age equivalent scores of cognitive testing measured from baseline (BSID-III or KABC-II) (Cohort A) | Baseline to Week 105
For regions other than US: Change in the age equivalent scores of adaptive behavior measured from baseline (VABS-II) (Cohort A) | Baseline to Week 105
For the US: Change in the raw scores of adaptive behavior measured from baseline (VABS-II) (Cohort A) | Baseline to Week 105
For all regions: Relative change in liver volume relative to body weight from baseline (Cohort A and Cohort B) | Baseline to Week 53
For all regions: Relative change in spleen volume relative to body weight from baseline (Cohort A and Cohort B) | Baseline to Week 53

CONTACTS AND LOCATIONS:
Locations (29):
- United States (7):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill Medical School Wing E, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hospital Universitario Austral, Buenos Aires, Argentina
- Brazil (3):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Instituto de Medicina Integral Prof. Fernando Figueira - Imip, Recife
  - Instituto de Genética e Erros Inatos do Metabolismo, São Paulo
- Fundación Cardio Infantil - Instituto de Cardiología, Bogotá, Colombia
- France (3):
  - Hôpital Femme Mère Enfant, Bron
  - Chu De Montpellier Hopital Gui De Chauliac, Montpellier
  - Hôpital Armand Trousseau, Paris
- Germany (4):
  - Universitätsklinikum Giessen, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - SphinCS GmbH, Höchheim
  - Universitätsmedizin Mainz, Mainz
- Israel (2):
  - Ha'Emek Medical Center, Afula
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (2):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Osp. Pediatrico Bambino Gesù, IRCCS, Rome
- Uniwersytecki Szpital Dziecięcy, Krakow, Poland
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- Turkey (Türkiye) (2):
  - Gazi University Medicine Faculty Hospital, Ankara
  - Ege University Children Hospital, Izmir
- Great Ormond Street Hospital for Children NHS Trust - Metabolic Medicine, London, United Kingdom